CLINICAL TRIAL: NCT02653014
Title: An Open-Label, Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KBP-5074 in Healthy Subjects With a Separate Panel in Subjects With Mild to Moderate Renal Impairment
Brief Title: Safety, Tolerability and Pharmacokinetics of KBP-5074 in Healthy Subjects and Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBP5074-1-002
Record Dates: First submitted 2015-12-29; First posted 2016-01-12 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — KBP-5074; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Healthy Volunteers will receive 2.5mg of KBP-5074, QD, 14 days
  Interventions: Drug: KBP-5074
- Cohort 2 (Experimental): Healthy Volunteers will receive 5.0mg of KBP-5074, QD, 14 days
  Interventions: Drug: KBP-5074
- Cohort 3 (Experimental): Subjects with mild to moderate renal impairment will receive 0.5mg of KBP-5074, QD, 56 days
  Interventions: Drug: KBP-5074
- Cohort 4 (Experimental): Subjects with mild to moderate renal impairment will receive 2.5mg of KBP-5074, QD, 56 days
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: KBP-5074
  Other Names: mineralocorticoid receptor antagonist

SUMMARY:
This multiple ascending dose (MAD) study in healthy subjects and subjects with mild to moderate renal impairment will evaluate the safety, tolerability and pharmacokinetics of KBP-5074. Safety/tolerability data and Pharmacokinetics (PK)/Pharmacodynamics (PD) (plasma aldosterone, serum potassium, UACR and Blood Pressure) relationships will be explored to support the selection of dosing regimens of KBP-5074 that are suitable for the Phase II/III study.

DETAILED DESCRIPTION:
This study consists of two parts: Part 1 is an open-label, multiple ascending dose (MAD) study to evaluate the safety, tolerability and pharmacokinetics of KBP-5074 in healthy subjects. The safety and tolerability will be assessed at each dose level before progressing to the next higher dose. Part 2 is an open label, randomized, parallel study to assess the safety and tolerability, the effect of renal dysfunction on the pharmacokinetics of KBP-5074, as well as the PK/PD relationship in subjects with mild to moderate renal impairment.

ELIGIBILITY:
Inclusion Criteria for Part 1:

* Healthy male or female subject
* Are between the ages of 18 and 45 years (inclusive);
* Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 50 kg.

Exclusion Criteria for Part 1:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
* Known or suspected malignancy;
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody;
* Positive pregnancy test result.

Inclusion Criteria for Part 2:

* Are between the ages of 18 and 75 years (inclusive);
* Mild to moderate chronic kidney disease (defined as estimated glomerular filtration rate (eGFR) > 30 and ≤89 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) formula, for > 3 months;
* Proteinuria (defined as urine albumin to creatinine ratio (UACR) ≥100 mg/g and ≤3,000 mg/g in two mid-morning urine specimens within a month interval);
* Subjects treated with an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)
* Serum potassium≥3.3 mmol/L and ≤4.8 mmol/L;
* Body mass index (BMI) of 19 to 40 kg/m2 inclusive and body weight not less than 50 kg.

Exclusion Criteria for Part 2:

* Severe uncontrolled hypertension (diastolic > 115 mmHg or systolic blood pressure > 180 mmHg) at either the Screening visit or the Study Check-in Visit;
* Type I diabetes mellitus or poorly controlled Type 2 diabetes mellitus (HbA1c > 10%) at the Screening visit;
* Prior kidney transplant, or anticipated need for transplant during study participation;
* Clinical diagnosis of heart failure and persistent symptoms (New York Heart Association [NYHA] Class II- IV) at either the Screening visit or the Study Check-in Visit;
* Known or suspected contraindications to study medications, including history of hypersensitivity or allergy to ACE inhibitors, ARBs, or aldosterone antagonists;
* Any clinically significant disorder, except for conditions associated with type 2 diabetes mellitus history, which in the investigators opinion could interfere with the results of the trial;
* Diabetic gastroparesis;
* Known bilateral clinically relevant renal artery stenosis (>75% reduction in artery diameter).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 69 days
  Rate of adverse events

SECONDARY OUTCOMES:
Area Under Curve (AUC) in healthy subjects | pre-dose and 2, 4, 6, 8, 10, 12, 18, and 24 hours post dose on Day 1; pre-dose on Days 8, 11, 12, and 13; and pre-dose and 2, 4, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 168, 216, 264, and 312 hours post dose on Day 14
  AUC 0-24 hours
Area Under Curve (AUC) in subjects with mild to moderate renal impairment | pre-dose and 2, 4, 6, 8, 10, 12, 18, and 24 hours post dose on Day 1; pre-dose on Days 8, 11, 12, and 13; pre-dose and 2, 4, 6, 8, 10, 12, 18, and 24 hours post dose on Day 14; pre-dose on Days 29 and 43; and pre-dose and 6, 12, and 24 hours on Day 56
  AUC 0-24 hours
The effect of mild to moderate renal impairment on the Area Under Curve (AUC) | Up to 15 days
  AUC 0-24 hours
Plasma aldosterone levels in healthy subjects | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Day 8; and 24 hours post last dose on Day 15
  Plasma aldosterone level
Serum potassium levels in healthy subjects | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Day 8; and 24 hours post last dose on Day 15
  Serum potassium level
Plasma aldosterone levels in subjects with mild to moderate renal impairment | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Days 8, 15, 29, and 43; and 24 hours post last dose on Day 57
  Plasma aldosterone level
Serum potassium levels in subjects with mild to moderate renal impairment | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Days 8, 15, 29, and 43; and 24 hours post last dose on Day 57
  Serum potassium level
Urinary Albumin to Creatinine Ratio (UACR) in subjects with mild to moderate renal impairment | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Days 8, 15, 29, and 43; and 24 hours post last dose on Day 57
  Ratio of urinary albumin level to creatinine level
Blood Pressure in subjects with mild to moderate renal impairment | Pre-dose, 6, and 24 hours post dose on Day 1; pre-dose on Days 8, 15, 29, and 43; and 24 hours post last dose on Day 57
  Systolic and diastolic seated blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Research by Design, LLC, Evergreen Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No